CLINICAL TRIAL: NCT03247673
Title: A Randomized, Double-blind, Three-arm, Parallel Group, Single-dose Study to Compare the Pharmacokinetics and Safety of Three Formulations of Bevacizumab (CT-P16, EU-approved Avastin and US-licensed Avastin) in Healthy Male Subjects
Brief Title: To Demonstrate Similarity of Pharmacokinetics and Evaluate Safety of CT-P16, EU-Approved Avastin and US-licensed Avastin
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Celltrion (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: CT-P16 1.1
Record Dates: First submitted 2017-08-03; First posted 2017-08-14 (Actual); Results first posted 2019-07-25 (Actual); Last update posted 2020-03-26 (Actual); Status verified 2020-03

CONDITIONS: Healthy
Keywords: safety; Pharmacokinetics; Immunogenicity
MeSH Terms: interventions — Bevacizumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- CT-P16 (Experimental): CT-P16 will be administrated once in IV infusion of 5mg/KG to healthy male subjects
  Interventions: Drug: CT-P16
- EU-approved Avastin (Active Comparator): EU-approved Avastin will be administrated once in IV infusion of 5mg/KG to healthy male subjects
  Interventions: Drug: EU-approved Avastin
- US-licensed Avastin (Active Comparator): US-licensed Avastin will be administrated once in IV infusion of 5mg/KG to healthy male subjects
  Interventions: Drug: US-licensed Avastin

INTERVENTIONS:
Drug: CT-P16 — CT-P16 is a biosimilar product for Avastin
  Other Names: bevacizumab
  Arms: CT-P16
Drug: EU-approved Avastin — EU-approved Avastin
  Other Names: bevacizumab
  Arms: EU-approved Avastin
Drug: US-licensed Avastin — US-licensed Avastin
  Other Names: bevacizumab
  Arms: US-licensed Avastin

SUMMARY:
This study is a Phase 1 Randomized, Double-blind, Three-arm, Parallel Group, Single-dose Study to compare the PK, safety and immunogenicity of the proposed biosimilar test product CT-P16 with EU-approved Avastin and US-licensed Avastin after a single IV infusion of 5mg/kg of each product to healthy male subjects

DETAILED DESCRIPTION:
This study is a double-blind, three-arm, parallel group, single-dose study. A total of 141 subjects will be enrolled; 47 subjects in each of the 3 arms of the clinical study. In each arm, all subjects will receive a single dose (5 mg/kg) of either CT-P16, EU-approved Avastin, or US-licensed Avastin by intravenous (IV) infusion for 90 min (±5 min) on Day 1 followed by 15 weeks during which the PK, safety, and immunogenicity measurements will be made. The randomization will be stratified by body weight and site.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male subjects between the ages of 19 and 55 years, both inclusive
* Body Mass Index (BMI) between 18.0 and 29.9 kg/m2 (both inclusive) and a body weight ≥ 50 kg

Exclusion Criteria:

* Subject is a female.
* Clinically significant allergic reactions, hypersensitivity
* A disease classed as significant by the Investigator
* Non-healing wound, ulcer, bone fracture, a major surgical procedure, significant traumatic injury
* Any malignancy
* Undergone treatment with an investigational drug or participated in another clinical trial
* Plans to father a child or donates sperms

Ages: 19 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 141 (Actual)
Dates: Start 2017-08-07 (Actual); Primary Completion 2017-12-22 (Actual); Study Completion 2018-01-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sung Young Lee, Study Director — Celltrion
Locations (3):
- South Korea (3):
  - Inje University Busan Paik Hospital, Busan
  - Inha University Hospital, Incheon
  - Seoul St.Mary's hospital, Seoul

REFERENCES:
- [Derived] Cho SH, Han S, Ghim JL, Nam MS, Yu S, Park T, Kim S, Bae J, Shin JG. A Randomized, Double-Blind Trial Comparing the Pharmacokinetics of CT-P16, a Candidate Bevacizumab Biosimilar, with its Reference Product in Healthy Adult Males. BioDrugs. 2019 Apr;33(2):173-181. doi: 10.1007/s40259-019-00340-x. PMID 30850957
- See also: Celltrion, Inc. homepage — http://www.celltrion.com

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | CT-P16 | EU-approved Avastin | US-licensed Avastin
Started | 46 | 47 | 48
Completed | 45 | 47 | 44
Not Completed | 1 | 0 | 4
Not completed — Withdrawal by Subject | 1 | 0 | 3
Not completed — Lost to Follow-up | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Safety Population
Groups:
- Total: Total of all reporting groups
Arm/Group | CT-P16 | EU-approved Avastin | US-licensed Avastin | Total
Number analyzed (Participants) | 46 | 47 | 48 | 141
Age, Continuous [Mean (Standard Deviation); unit: years] | 28.5 (8.69) | 28.4 (7.59) | 26.5 (6.28) | 27.8 (7.57)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0
  Male | 46 | 47 | 48 | 141
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 46 | 47 | 48 | 141
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 0 | 0 | 0 | 0
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  South Korea | 46 | 47 | 48 | 141
Weight (kg) [Mean (Standard Deviation); unit: kg] | 69.93 (9.073) | 71.01 (9.417) | 69.54 (8.141) | 70.16 (8.845)
BMI [Mean (Standard Deviation); unit: kg/m^2] — kg/m2
  kg/m^2 | 22.89 (2.310) | 23.20 (2.492) | 23.17 (2.303) | 23.09 (2.357)

OUTCOME MEASURES:

1. Primary Outcome: AUC0-inf
Description: Area under the concentration-time curve from time zero to infinity
Time Frame: pre-dose, end of infusion, 1 hour after EOI, 4, 8, 12, 24, 48, 72, 168, 336, 672, 1,008, 1,344, 1,680, 2,016, and 2,352 hours after SOI
Population: PK population
Measure: Mean (Standard Deviation); unit: h*ug/mL
Arm/Group | CT-P16 | EU-approved Avastin | US-licensed Avastin
Number analyzed (Participants) | 46 | 47 | 48
h*ug/mL | 42034.90 (6070.668) | 40413.44 (5012.778) | 43017.95 (5782.951)

2. Primary Outcome: Cmax
Description: Maximum Serum Concentration (Cmax)
Time Frame: as for outcome 1
Population: PK population
Measure: Mean (Standard Deviation); unit: ug/mL
Arm/Group | CT-P16 | EU-approved Avastin | US-licensed Avastin
Number analyzed (Participants) | 46 | 47 | 48
ug/mL | 117.22 (17.756) | 114.06 (15.391) | 113.09 (17.402)

3. Primary Outcome: AUC0-last
Description: Area Under the Concentration-time Curve From Time Zero to the Last Quantifiable Concentration
Time Frame: as for outcome 1
Population: PK population
Measure: Mean (Standard Deviation); unit: h*ug/mL
Arm/Group | CT-P16 | EU-approved Avastin | US-licensed Avastin
Number analyzed (Participants) | 46 | 47 | 48
h*ug/mL | 41142.81 (5694.184) | 39411.98 (4649.319) | 41804.05 (5463.814)

4. Secondary Outcome: Additional Pharmacokinetics (Time to Cmax)
Description: To assess the additional PK of study drugs (Time to Cmax)
Time Frame: as for outcome 1
Population: PK population
Measure: Median (Full Range); unit: h
Arm/Group | CT-P16 | EU-approved Avastin | US-licensed Avastin
Number analyzed (Participants) | 46 | 47 | 48
h | 2.5 [1.5 to 12.0] | 2.5 [1.5 to 8.0] | 2.5 [1.5 to 8.0]

5. Secondary Outcome: Number of Participants With Anti-Drug Antibody Positive
Description: number of participants with anti-drug antibody positive at post-dose
Time Frame: up to 15 weeks
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | CT-P16 | EU-approved Avastin | US-licensed Avastin
Number analyzed (Participants) | 46 | 47 | 48
Participants | 2 | 2 | 3

ADVERSE EVENTS:
Time Frame: up to 15 weeks
Arm/Group | CT-P16 | EU-approved Avastin | US-licensed Avastin
All-Cause Mortality (participants affected / at risk) | 0/46 | 0/47 | 0/48
Serious Adverse Events (participants affected / at risk) | 0/46 | 0/47 | 0/48
Other Adverse Events (participants affected / at risk) | 15/46 | 22/47 | 17/48
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | CT-P16 (N=46) | EU-approved Avastin (N=47) | US-licensed Avastin (N=48)
Diarrhea (Gastrointestinal disorders) | 3 | 6 | 4
Nasopharyngitis (Infections and infestations) | 4 | 1 | 6
Blood creatine phosphokinase increased (Investigations) | 3 | 5 | 4
C-reactive protein increased (Investigations) | 2 | 5 | 4
Infusion-related reaction (Injury, poisoning and procedural complications) | 2 | 2 | 4
Headache (Nervous system disorders) | 1 | 2 | 3
Troponin I increased (Investigations) | 1 | 3 | 0
White blood cell count decreased (Investigations) | 1 | 0 | 3

LIMITATIONS AND CAVEATS:
Subject with unreliable PK parameter results were excluded from summary. Only treatment-emergent adverse events were summarized.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (2):
  • Statistical Analysis Plan (2018-03-29): https://cdn.clinicaltrials.gov/large-docs/73/NCT03247673/SAP_002.pdf
  • Study Protocol (2017-06-07): https://cdn.clinicaltrials.gov/large-docs/73/NCT03247673/Prot_003.pdf